CLINICAL TRIAL: NCT02479763
Title: A Randomized Comparison Between Conventional and Waveform-Confirmed Loss-of-Resistance for Thoracic Epidural Blocks
Brief Title: A Comparison Between Conventional and Waveform-Confirmed Loss-of-Resistance for Thoracic Epidural Blocks
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Montreal General Hospital (Other)
Responsible Party: Principal Investigator, De QH Tran, Associate professor, Montreal General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-077 MUHC
Record Dates: First submitted 2015-06-22; First posted 2015-06-24 (Estimated); Results first posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-01

CONDITIONS: Anesthesia
Keywords: Epidural waveform analysis; Loss of resistance

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional loss-of-resistance (No Intervention)
- Waveform-confirmed loss-of-resistance (Experimental)
  Interventions: Procedure: Waveform-confirmed loss-of-resistance

INTERVENTIONS:
Procedure: Waveform-confirmed loss-of-resistance — Using waveform analysis to confirm thoracic epidural space
  Arms: Waveform-confirmed loss-of-resistance

SUMMARY:
In the investigators' institution, the failure rate for thoracic epidural blocks is 23.1%. This stems from the prevalence of trainee operators coupled with the non-specific nature of loss-of-resistance. In the current randomized trial, we will set out to compare conventional and epidural waveform analysis-confirmed loss-of-resistance. The investigators' research hypothesis is that loss-of-resistance combined with epidural waveform analysis will decrease the failure rate of thoracic epidural blocks.

ELIGIBILITY:
Inclusion Criteria:

* the patients undergoing thoracic epidural catheter insertion for thoracic and abdominal surgery or rib fractures with American Society of Anesthesiologists (ASA) classification 1-3 and body mass index between 18 and 35

Exclusion Criteria:

* adults who are unable to give their own consent
* coagulopathy (assessed by history and physical examination and, if deemed clinically necessary, by blood work up ie platelets ≤ 100, or International Normalized Ratio ≥ 1.4)
* renal failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up ie creatinine ≥ 100)
* hepatic failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up ie transaminases ≥ 100)
* allergy to local anesthetic (LA)
* pregnancy
* prior surgery in the thoracic spine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: De QH Tran, Principal Investigator — McGill University
Locations (2):
- Montreal General Hospital, McGill University, Montreal, Quebec, Canada
- Ramathibodi Hospital, Mahidol University, Ratchathewi, Bangkok, Thailand

RESULTS

PARTICIPANT FLOW:
Groups:
- Conventional Loss-of-resistance: Conventional loss-of-resistance: Using tactile feeling to identify thoracic epidural space
Period: Overall Study
Arm/Group | Conventional Loss-of-resistance | Waveform-confirmed Loss-of-resistance
Started | 53 | 53
Completed | 50 | 50
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Loss-of-resistance | Waveform-confirmed Loss-of-resistance | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (11.0) | 61.1 (11.8) | 61.3 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 20 | 36
  Male | 34 | 30 | 64
BMI (kg/m^2), Continuous [Mean (Standard Deviation); unit: kg/m^2] | 25.5 (4.4) | 24.6 (3.7) | 25.1 (4.1)
American Society of Anesthesiologists (ASA) physical status, Categorical [Number; unit: participants] — The ASA physical status classification system is a system for assessing the fitness of patients before surgery. There are six classes depending on status of patients. While ASA class I is a normal healthy patient, ASA class VI is a declared brain-dead patient.
  participants
    Class I; A normal healthy patient | 3 | 9 | 12
    Class II; A patient with mild systemic disease | 21 | 23 | 44
    Class III; A patient with severe systemic disease | 26 | 18 | 44

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Successful Epidural Blocks
Description: Fifteen minutes after the LA injection, a blinded observer will apply ice to the T1-L4 dermatomes and assess the epidural block. The criterion standard for success will be the presence of an epidural block (defined as a block to ice in at least 2 dermatomes bilaterally). If the operators cannot thread the catheter after 2 attempts, epidural blocks will considered failures.
Time Frame: up to 15 minutes after the procedure
Measure: Number; unit: percentage of patients
Arm/Group | Conventional Loss-of-resistance | Waveform-confirmed Loss-of-resistance
Number analyzed (Participants) | 50 | 50
percentage of patients | 76 | 98

ADVERSE EVENTS:
Arm/Group | Conventional Loss-of-resistance | Waveform-confirmed Loss-of-resistance
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 2/50 | 2/50
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Loss-of-resistance (N=50) | Waveform-confirmed Loss-of-resistance (N=50)
Transient self-resolving paresthesia (Nervous system disorders) | 0 (0) | 2 (2)
Vascular breach (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No